CLINICAL TRIAL: NCT01735123
Title: Early Dietary Intervention and Later Signs of Beta-Cell Autoimmunity: Potential Mechanisms
Brief Title: Early Dietary Intervention and Later Signs of Beta-Cell Autoimmunity
Acronym: EDIA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Helsinki (Other)
Collaborators: University of Turku (Other); Finnish Institute for Health and Welfare (Other Government); Tampere University Hospital (Other)
Responsible Party: Principal Investigator, Mikael Knip, Professor, University of Helsinki
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 1DP3DK094338-01 (NIH)
Record Dates: First submitted 2012-11-24; First posted 2012-11-28 (Estimated); Last update posted 2017-02-27 (Actual); Status verified 2017-02

CONDITIONS: Diabetes Mellitus, Type 1
Keywords: infant formula; diet; diabetes mellitus, type 1; autoimmunity
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Autoimmune Diseases | interventions — Diet Therapy

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- extensively hydrolyzed casein formula (Experimental): The investigators plan to randomize 60 out of 120 infants to be weaned to an extensively hydrolyzed casein formula. Recruited mothers are encouraged to breast-feed. The dietary intervention will be applied until 9 months of age. The minimum exposure time to the study formula should be 90 days. Signs of beta-cell autoimmunity, i.e. diabetes-associated autoantibodies, will be monitored in the study participants, although the study will not have sufficient power to detect statistically significant differences in the seroconversion rate between the groups due to the limited number of infants randomized.
  Interventions: Dietary Supplement: dietary intervention
- cow's milk based infant formula (Experimental): The investigators plan to randomize 60 out of 120 infants to be weaned to a cow's milk based infant formula. Recruited mothers are encouraged to breast-feed. The dietary intervention will be applied until 9 months of age. The minimum exposure time to the study formula should be 90 days. Signs of beta-cell autoimmunity, i.e. diabetes-associated autoantibodies, will be monitored in the study participants, although the study will not have sufficient power to detect statistically significant differences in the seroconversion rate between the groups due to the limited number of infants randomized.
  Interventions: Dietary Supplement: dietary intervention

INTERVENTIONS:
Dietary Supplement: dietary intervention — hydrolyzed vs. nonhydrolyzed infant formula
  Other Names: An extensively hydrolyzed casein formula; A regular cow's milk based formula

SUMMARY:
The proposed mechanistic formula feeding study sets out to identify the mechanism(s) by which an extensively hydrolyzed casein formula is able to protect children at risk for type 1 diabetes (T1D) from beta-cell autoimmunity.

DETAILED DESCRIPTION:
Based on clinical and experimental observations the study will focus on defining the effects of two different formulas on intestinal permeability, IL (interleukin)-17 immunity, serum metabolome, and gut microflora. The study will be based on a randomized pilot intervention trial using an intention to treat statistical analysis to compare e.g. gut permeability between the two treatment groups. The investigators hypothesize that the extensively hydrolyzed casein formula decreases intestinal permeability, down-regulates IL-17 immunity and proinflammatory lysophosphatidylcholines, and stabilize Lactobacilli levels in the gut microflora when compared to the conventional cow's milk formula. The study population comprises 120 newborn infants with HLA(Human Leukocyte Antigen)-conferred susceptibility to T1D. The mothers will be encouraged to exclusively breast-feed their infants as long as possible. The timing of weaning and introduction of study formula will be left to the mother. The infants are randomized to be weaned to one of two study formulas: ( i) standard cow's milk formula and (ii) an extensively hydrolyzed casein formula. The target will be that the infant should be exposed to his/her study formula for at least 90 days before the age of 270 days. The diet of the infant will be studied with 3-day food records at the age of 3, 6, 9, and 12 months of age. To estimate the amount of breast milk received the weight of the infant will be measured just before and after each lactation. The HLA genotype will be analyzed from cord blood, and the result will be available within 10 days after birth. The family will visit the Study Center when the infant is 3, 6, 9, and 12-month-old. Blood samples will be obtained on each visit. In addition the families are asked to collect stool samples at home once a month during the study. Intestinal permeability will be assessed with the lactulose/mannitol test at the age of 3, 6, 9, and 12 months. Gut microflora will be analyzed with high-throughput, culture-independent methods and serum metabolome with established metabolomics platforms. Il-17 immunity will be studied using peripheral blood mononuclear cells. This work will generate novel knowledge of the disease process leading to overt T1D by studying potential mechanism(s) mediating the protective effect conferred by an extensively hydrolyzed casein formula against beta-cell autoimmunity. The identification of such mechanism(s) will most likely facilitate the refinement of effective preventive measures based on modifications of early infant nutrition.

ELIGIBILITY:
Inclusion Criteria:

- The infant's parents give signed consent to participate and their HLA genotype is eligible.

Exclusion Criteria:

* An older sibling of the newborn infant has been included in this study;
* Multiple gestation;
* The parents are unwilling or unable to feed the infant cow's milk based products for any reason (e.g., religious, cultural);
* The gestational age of the newborn infant is less than 35 weeks
* Inability of the family to take part in the study (e.g. the family had no access to the Study Center or telephone)
* The newborn infant has a recognizable severe illness such as those due to chromosomal abnormality, congenital malformation, respiratory failure needing assisted ventilation, enzyme deficiencies, etc.;
* The infant receives any infant formula other than study formula or Nutramigen at the delivery hospital
* No HLA sample has been drawn before the age of 8 days.

Max Age: 12 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 87 (Actual)
Dates: Start 2013-01; Primary Completion 2016-07 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
Intestinal permeability will be determined at the age of 3, 6, 9 and 12 months with the lactulose/mannitol test Intestinal permeability at the age of 9 months assessed with the lactulose/mannitol test | 3, 6, 9 and 12 months
  Intestinal permeability will be determined at the age of 3, 6, 9 and 12 months with the lactulose/mannitol test

SECONDARY OUTCOMES:
Serum metabolic profile | 3, 6, 9 and 12 months
  The serum metabolic profile wil be analyzed with metabolomics at the age of 3, 6, 9, and 12 months

OTHER OUTCOMES:
Intestinal microbiome | 3, 6, 9 and 12 months
  The intestinal microbiome will be analyzed at the age of 3, 6, 9 , and 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Mikael Knip, M.D., Principal Investigator — University of Helsinki
Locations (1):
- Tampere University Hospital, Tampere, Finland

REFERENCES:
- [Derived] Lalli MK, Salo TE, Hakola L, Knip M, Virtanen SM, Vatanen T. Associations between dietary fibers and gut microbiome composition in the EDIA longitudinal infant cohort. Am J Clin Nutr. 2025 Jan;121(1):83-99. doi: 10.1016/j.ajcnut.2024.11.011. Epub 2024 Nov 16. PMID 39551356
- [Derived] Koivusaari K, Niinisto S, Nevalainen J, Honkanen J, Ruohtula T, Koreasalo M, Ahonen S, Akerlund M, Tapanainen H, Siljander H, Miettinen ME, Alatossava T, Ilonen J, Vaarala O, Knip M, Virtanen SM. Infant Feeding, Gut Permeability, and Gut Inflammation Markers. J Pediatr Gastroenterol Nutr. 2023 Jun 1;76(6):822-829. doi: 10.1097/MPG.0000000000003756. Epub 2023 Mar 12. PMID 36913717
- [Derived] Lamichhane S, Siljander H, Salonen M, Ruohtula T, Virtanen SM, Ilonen J, Hyotylainen T, Knip M, Oresic M. Impact of Extensively Hydrolyzed Infant Formula on Circulating Lipids During Early Life. Front Nutr. 2022 May 24;9:859627. doi: 10.3389/fnut.2022.859627. eCollection 2022. PMID 35685890
- [Derived] Siljander H, Jason E, Ruohtula T, Selvenius J, Koivusaari K, Salonen M, Ahonen S, Honkanen J, Ilonen J, Vaarala O, Virtanen SM, Lahdeaho ML, Knip M. Effect of Early Feeding on Intestinal Permeability and Inflammation Markers in Infants with Genetic Susceptibility to Type 1 Diabetes: A Randomized Clinical Trial. J Pediatr. 2021 Nov;238:305-311.e3. doi: 10.1016/j.jpeds.2021.07.042. Epub 2021 Jul 20. PMID 34293372